CLINICAL TRIAL: NCT00877487
Title: A Phase 4, Double-Blind, Multi-Center, Placebo-Controlled, Randomized Withdrawal, Safety and Efficacy Study of SPD489 in Adults Aged 18-55 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy of Vyvanse in Adults With Attention-Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-401
Record Dates: First submitted 2009-03-19; First posted 2009-04-07 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SPD489 (Experimental)
  Interventions: Drug: SPD489 (Lisdexamfetamine dimesylate)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD489 (Lisdexamfetamine dimesylate) — 1 capsule (either 30, 50, or 70mg strength) per day for 6 weeks.
  Other Names: Vyvanse
  Arms: SPD489
Drug: Placebo — 1 capsule (identical to drug capsules) per day for 4 weeks during the double blind period.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the maintenance of efficacy, as measured by Adult ADHD Rating Scale with Prompts (Adult ADHD-RS with prompts) and Clinical Global Impression - Severity (CGI-S) scores, through a randomized withdrawal design when subjects with ADHD have been on stable treatment with commercial SPD489 for a minimum of 6 months and are maintained on their screening dose of commercial SPD489.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18-55 years of age, inclusive at the time of consent.
2. Female subjects must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test at Screening and a negative urine pregnancy test at baseline and agree to comply with any applicable contraceptive requirements of the protocol.
3. Subject has a documented diagnosis of ADHD or meets DSM-IV-TR™ with adult prompts criteria by history for a primary diagnosis of ADHD prior to treatment.
4. Subject has a Baseline score of <22 using the Adult ADHD-RS with prompts and CGI-S score ≤3.
5. Subject has been on stable treatment with commercial SPD489 (30, 50, or 70mg) for a minimum of at least 6 months preceding the Screening Visit with acceptable tolerability.Prior treatment with commercial SPD489 in the 6 months preceding the Screening Visit must be documented by prescription records, prescribing physician notes, or pharmacy records. Those subjects whose primary care physician (PCP) is someone other than the Principal Investigator (PI) will be required to provide the above documentation to the site.
6. Subject must have a minimum level of intellectual functioning, as determined by the Investigator.
7. Subject is willing and able to comply with all the testing and requirements defined in this protocol.
8. Subject is able to swallow a capsule.
9. Subject must be able to provide written, personally signed and dated informed consent to participate in the study, in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E627 and applicable regulations, before completing any study-related procedures.

Exclusion Criteria:

1. Subject has a current comorbid psychiatric disorder that is either controlled with medications prohibited in this study or is uncontrolled and associated with significant symptoms. Prohibited disorders include those associated with diagnoses including but not limited to any severe comorbid Axis II disorder or severe Axis I disorder (such as Post Traumatic Stress Disorder [PTSD], psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder). Other symptomatic manifestations (such as agitated states)that contraindicate treatment with SPD489 or confound efficacy or safety assessments in the opinion of the examining physician are also prohibited. Comorbid psychiatric diagnoses will be established by the psychiatric evaluation that includes the Structured Clinical Interview for DSM-IV-TR™ disorders (SCID-I).
2. Subject is currently considered a suicide risk, has previously made a suicide attempt or has a prior history of, or is currently demonstrating suicidal ideation.
3. The subject has a body mass index (BMI) of <18.5 or ≥40.
4. Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments administered in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional condition(s) that in the Investigator's opinion would prohibit the subject from completing the study or would not be in the best interest of the subject. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol. Mild, stable asthma is not exclusionary.
5. Subject has a history of seizures (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder.
6. Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, transient ischemic attack or stroke or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
7. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
8. Subject has any clinically significant ECG or clinically significant laboratory abnormality at Screening.
9. Subject has current abnormal thyroid function, as defined as abnormal Screening thyroid stimulating hormone (TSH) and thyroxine (T4). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
10. Subject has a history of moderate to severe hypertension or has a resting sitting systolic blood pressure >139mmHg or diastolic blood pressure >89mmHg. Subjects with well-controlled mild or moderate hypertension on a single antihypertensive agent are allowed.
11. Subject is taking any medication that is excluded (Please refer to Table 2).
12. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamines.
13. Subject has a recent history (within the past 6 months) of suspected substance abuse or dependence disorder (excluding nicotine) in accordance with DSM-IV-TR™ criteria.
14. Subject has a positive urine drug result at Screening (with the exception of subject's current stimulant therapy).
15. Subject has taken an investigational compound that has a central nervous system(CNS) effect or taken part in a clinical trial for ADHD 6 months prior to the Screening Visit.
16. Subject has taken part in an investigational trial within the 30 days prior to the Screening Visit.
17. Subject has glaucoma.
18. Subject is taking other medications that have CNS effects or affect performance, such as chronic use of sedating antihistamines and decongestant sympathomimetics (7 days prior to Screening). Stable use of bronchodilator inhalers is not exclusionary.
19. Subject is female and pregnant or lactating.
20. Subjects who have previously been enrolled into this study and subsequently withdrawn.
21. Subject is not well controlled on SPD489 with acceptable tolerability (Adult ADHD-RS with prompts score ≥22).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2010-07-08 (Actual); Study Completion 2010-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (55):
- United States (55):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Valley Clinical Research, Inc., El Centro, California
  - Peninsula Research Associates, Inc, Rolling Hills Estates, California
  - PCSD Feighner Research, San Diego, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Colorado Clinica Trials, Inc., Highlands Ranch, Colorado
  - Florida Clinical Research Center, Bradenton, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Fidelity Clinical Research, Inc., Lauderhill, Florida
  - CNS Healthcare, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Joliet Center for Clinical Research, Joliet, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - CIENTIFICA, Inc, Newton, Kansas
  - Psychiatric Associates, Overland Park, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Clinical Trial Technology Inc., Prairie Village, Kansas
  - Pedia Research LLC, Owensboro, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Rockville, Maryland
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - The Behavioral Medicine Clinic of NW Michigan, Traverse City, Michigan
  - Behavioral Medical Center-Troy, Troy, Michigan
  - Midwest Research Group/ St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Global Medical Institutes, LLC. Princeton Medical Institute, Princeton, New Jersey
  - Richmond Behavioral Associates, Staten Island, New York
  - Richard H. Weisler, MD, PA & Associates, Raleigh, North Carolina
  - Prarie St. Johns/ Odyssey Research, Fargo, North Dakota
  - UHCMC/ Discovery and Wellness Center for Children, Cleveland, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Calcagno Pediatrics, Gresham, Oregon
  - Introspect of Buxmont, Ltd., Colmar, Pennsylvania
  - Youth and Family Research Program, Pittsburgh, Pennsylvania
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - CNS Healthcare, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Bayou City Reserch, Ltd., Houston, Texas
  - Westex Clinical Investigators, Lubbock, Texas
  - Cerebral Research, LLC, San Antonio, Texas
  - Aspen Clinical Research, Orem, Utah
  - Vermont Clinical Study Center, Burlington, Vermont
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Psychiatric Alliance of the Blue Ridge, Charlottesville, Virginia
  - Dominion Clinical Research, Midlothian, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Dean Foundation, Middleton, Wisconsin

REFERENCES:
- [Result] Brams M, Weisler R, Findling RL, Gasior M, Hamdani M, Ferreira-Cornwell MC, Squires L. Maintenance of efficacy of lisdexamfetamine dimesylate in adults with attention-deficit/hyperactivity disorder: randomized withdrawal design. J Clin Psychiatry. 2012 Jul;73(7):977-83. doi: 10.4088/JCP.11m07430. Epub 2012 Jun 12. PMID 22780921
- [Derived] Weisler RH, Babcock T, Adeyi B, Brams M. Relationship of ADHD symptoms and global illness severity in adults treated with lisdexamfetamine dimesylate. Postgrad Med. 2014 Sep;126(5):31-41. doi: 10.3810/pgm.2014.09.2798. PMID 25295648
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects had been on stable treatment with commercial SPD489 (30, 50, or 70 mg/day) for at least 6 months. They then entered a 3-week open-label treatment phase on SPD489 (30, 50, or 70 mg/day). They then entered a 6-week double-blind randomized withdrawal phase where they were assigned to either SPD489 or placebo treatment group.
Groups:
- SPD489: Subjects receive SPD489 at 30, 50, or 70 mg/day.
- Placebo: Subjects who previously were receiving SPD489 are now only getting placebo.
Period: Open-label Treatment Phase
Arm/Group | SPD489 | Placebo
Started | 123 | 0
Completed | 116 | 0
Not Completed | 7 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Out of country for business | 1 | 0
Period: Double-blind Randomized Withdrawal Phase
Arm/Group | SPD489 | Placebo
Started | 56 | 60
Completed | 50 | 13
Not Completed | 6 | 47
Not completed — Relapse criteria met | 5 | 45
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Moved out of state | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | SPD489
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (11.16)
Age, Customized [Count of Participants; unit: Participants] — The demographics are based on the safety population defined as all subjects who entered the open-label treatment phase and took at least 1 dose of investigational product (SPD489). 123 subjects enrolled into the study, but 1 subject withdrew prior to receiving a dose of investigational product in the open-label treatment phase. Therefore, 122 subjects are in the safety population.
  Participants
    Between 18 and 55 years | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 54
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 122

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) With Adult Prompts Total Score at up to 6 Weeks
Description: The ADHD-RS consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Up to 6 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 56 | 60
Units on a scale | 1.6 (1.39) | 16.8 (1.35)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -15.23, 95% CI 2-sided [-19.1 to -11.4]

2. Secondary Outcome: Assessment of Clinical Global Impression-Severity of Illness (CGI-S) at up to 6 Weeks
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: Up to 6 weeks
Population: FAS
Measure: Number; unit: Percent of Participants
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 56 | 60
Percent of Participants
  Normal, not at all ill | 32.1 | 5.0
  Borderline mentally ill | 35.7 | 11.7
  Mildly ill | 17.9 | 11.7
  Moderately ill | 7.1 | 33.3
  Markedly ill | 7.1 | 35.0
  Severely ill | 0 | 3.3
  Among the most extremely ill | 0 | 0
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

3. Primary Outcome: Percent of Treatment Failures at up to 6 Weeks
Description: Treatment failure defined as > or equal to 50% increase in the ADHD-RS with adult prompts total score and a > or equal to 2 point increase in the CGI-S score.
Time Frame: Up to 6 weeks
Population: Full Analysis Set (FAS) defined as all subjects who were randomized and received at least 1 dose of investigational product.
Measure: Number; unit: Percent of participants
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 56 | 60
Percent of participants | 8.9 | 75.0
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared

ADVERSE EVENTS:
Description: Safety Population defined as all subjects who entered the open-label treatment phase and took at least 1 dose of investigational product (SPD489).
Arm/Group | SPD489 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/56 | 1/60
Other Adverse Events (participants affected / at risk) | 16/56 | 6/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD489 (N=56) | Placebo (N=60)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD489 (N=56) | Placebo (N=60)
Headache (Nervous system disorders) | 8 (8) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.